CLINICAL TRIAL: NCT05683678
Title: US Selumetinib Registry
Status: Terminated | Type: Observational
Why Stopped: Sponsor decision.
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: ALX-NF1-501
Record Dates: First submitted 2023-01-05; First posted 2023-01-13 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-03

CONDITIONS: Neurofibromatosis Type 1; Plexiform Neurofibromas
Keywords: neurofibromatosis type 1; plexiform neurofibromas; NF1; PNs
MeSH Terms: conditions — Neurofibromatosis 1; Neurofibroma, Plexiform

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Cohort 1: Participants who started selumetinib and discontinued selumetinib before enrollment (the "discontinued" cohort).
- Cohort 2: Participants who started selumetinib before enrollment and are continuing to receive selumetinib at the time of enrollment (the "continuing" cohort).
- Cohort 3: Participants who started selumetinib on the day of enrollment or intend to initiate selumetinib within 3 months after enrollment (the "initiating" cohort).

SUMMARY:
The purpose of this study is to understand treatment patterns and assess long-term effectiveness and safety outcomes associated with selumetinib treatment as well as to explore clinical and non-clinical factors affecting those outcomes in patients with neurofibromatosis type 1 (NF1) and plexiform neurofibromas (PNs) who started selumetinib between the ages of 2 to 18 years inclusive, and initiated selumetinib treatment on or after 10 April 2020 in a real-world setting.

DETAILED DESCRIPTION:
This is a US observational registry of pediatric NF1 PN participants treated with selumetinib.

ELIGIBILITY:
Inclusion Criteria:

* Participants diagnosed with NF1 and PN
* Started selumetinib between the ages of 2 to 18 years inclusive, and initiated selumetinib treatment on or after 10 April 2020, including patients who:
* Discontinued selumetinib before enrollment; or
* Initiated treatment before enrollment and are currently on selumetinib; or
* Initiated selumetinib on the day of enrollment or intend to initiate selumetinib within 3 months after enrollment
* Able to give written informed consent. Participant or participant's parent/legal guardian must be willing and able to give written informed consent and the participant (if minor) must be willing to give written informed assent.

Exclusion Criteria:

* Participants currently participating in any clinical trials at time of enrollment or initiation of selumetinib.

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Approximately 200 participants who meet the eligibility criteria will be enrolled from 20-25 sites.
Sampling Method: Non-Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2019-01-04 (Actual); Primary Completion 2024-11-13 (Actual); Study Completion 2024-11-13 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Improvement in Clinically Significant Plexiform Neurofibromas (PNs) as Assessed by the Treating Physician | Up to Month 60
Number of Participants with Improvement in Disease Status as Assessed by the Treating Physician | Up to Month 60
Number of Participants with Improvement in Neurofibromatosis type 1 (NF1) Skeletal Manifestations | Up to Month 60
  Skeletal manifestations may include changes in the angle of spine curvature.
Number of Participants with Treatment Emergent Medical Events of Interest (MEOI) | Up to Month 60

SECONDARY OUTCOMES:
Change From Baseline in the Numerical Rating Scale (NRS-11) Score at Month 60 | Baseline, Month 60
Change From Baseline in the Pain Interference Index (PII) Score at Month 60 | Baseline, Month 60
Change From Baseline in the Patient Global Impression of Change (GIC) Scale at Month 60 | Baseline, Month 60
Change From Baseline in the Pediatric Quality of Life Inventory (PedsQL) at Month 60 | Baseline, Month 60

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Children's Hospital Los Angeles, Los Angeles, California
  - Nicklaus Children's Hospital, Miami, Florida
  - Arnold Palmer Hospital For Children, Orlando, Florida
  - Ochsner Medical Center, New Orleans, Louisiana
  - Mayo Clinic, Rochester, Minnesota
  - Albany Medical Center, Albany, New York
  - Waters Center for Childrens Cancer and Blood Disorders, Syracuse, New York
  - The Children's Hospital at Montefiore (CHAM), The Bronx, New York
  - Cook Children's Medical Center, Fort Worth, Texas

IPD SHARING:
Plan to Share IPD: Yes
Alexion has a public commitment to allow requests for access to study data and will be supplying a protocol, CSR, and plain language summaries.
Supporting Information: Study Protocol, SAP, CSR